CLINICAL TRIAL: NCT06899451
Title: Impact of Basophobia on Balance and Functional Outcomes in Patients With Stroke.
Acronym: stroke
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: AlRyada University for Science & Technology (Other)
Responsible Party: Principal Investigator, Heba Mohamed Gaber, Physical Therapy for Neuromuscular Disorders , Faculty of Physical Therapy, Cairo University
Other Study IDs: PT.BU.EC.13
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Balance
Keywords: fear of falling, balance, stroke
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- basophobia in stroke patients: The study will be conducted on 80 stroke patients , will randomly assigned to one of two groups using a secure system of opaque closed envelopes as study group (GA) and control group (GB) : -
  -
  Interventions: Other: systematic desensitization and balance

INTERVENTIONS:
Other: systematic desensitization and balance — 1. Systematic desensitization: 2 techniques
     1. Jacobson's technique (progressive muscle relaxation):
     2. Guided imagery training is a relaxation technique
  2. Goal-directed paradigm (selected program)
  Other Names: goal directed paradigm and balance

SUMMARY:
Several studies have reported that the physical functions associated with falls, including motor performance, postural balance, flexibility, and muscle strength, are also associated with FoF. Patients with stroke have trouble performing ADLs, including washing their face, eating, bathing, dressing, toileting, and walking, which also affect FoF. Anxiety and depression are common affective disorders in patients with stroke and significantly increase FoF .

DETAILED DESCRIPTION:
People who are afraid of falling because they can't keep their balance can utilize This makes them less susceptible to fall and high tendency to prevent it.

ELIGIBILITY:
Inclusion Criteria:

an ischemic stroke and having had the disease for longer than three months have frequent falling, having sufficient cognition (as measured by a Montreal Cognitive Assessment score of over 26) and having upper and lower extremity spasticity ranging from (grade 1+: 2) on a modified Ashworth scale

Exclusion Criteria

) Musculoskeletal issues, such as severe arthritis, total hip arthroplasty, knee surgery, lower extremity fractures within the previous six months, or contractures brought on by a fixed deformity and/or disparity in leg length, 2) Instable medical conditions (e.g., unstable angina, recent myocardial infarction, history of congestive heart failure, major heart valve problems, or unstable hypertension);

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with stroke
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 5 months
  is a five-point scaling score, a range of Zero - 4. "Zero" was given at the least level of function, while grade "4" will be given at the highest level of function. The scores are classified as follows: 41-56 = low fall risk, 21-40 = medium fall risk, and 0 -20 = high fall risk
The 16-item Fall Efficacy Scale-International | 5 months
  utilized to evaluate fear of falls.Varying from one (not concerned) to four (very concerned). For data analysis, the overall score, which was the sum of the 16 answers and ranged from 16 to 64 points, was utilized. A greater total score means the patients are more concerned about falling
Timed Up and Go Test (TUG) | 5 months
  starts with the patient getting up from the chair, walk 3 meters once a signal is given, walk 3 meters back to the chair, and then sit down calculating time taken by the patient

SECONDARY OUTCOMES:
fear of falling | 5 months
  Biodex Balance Systems

CONTACTS AND LOCATIONS:
Overall Officials: Heba Gaber, phd, Study Chair — ALRyada university for science and technology
Locations (1):
- Cairou, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.